CLINICAL TRIAL: NCT03952169
Title: Role of Probiotics in the Management of Hypercholesterolemia
Brief Title: Effect of Probiotics on Lipid Management
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Min Xia, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ProHealth-1
Record Dates: First submitted 2019-05-12; First posted 2019-05-16 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Primary Hypercholesterolemia
Keywords: Primary Hypercholesterolemia; Probiotics; Cardiovascular risk

STUDY DESIGN:
Intervention Model Description: placebo-controlled, randomized clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, investigators and care providers at the scene are all blinded to the allocation of treatment group. Data collected will be analyzed by another investigator who is blinded to the study design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics group (Experimental): Participants will be given capsules containing Lactobacillus paracasei once daily for 12 weeks followed by comprehensive physical and clinical examinations.
  Interventions: Dietary Supplement: Lactobacillus paracasei dietary supplement
- Placebo group (Placebo Comparator): Participants will be given capsules containing microcrystalline cellulose once daily for 12 weeks followed by comprehensive physical and clinical examinations.
  Interventions: Other: Placebo controls

INTERVENTIONS:
Dietary Supplement: Lactobacillus paracasei dietary supplement — a commercial probiotic dietary supplement
  Arms: Probiotics group
Other: Placebo controls — placebo with a similar appearance to probiotics supplement
  Arms: Placebo group

SUMMARY:
Dysbiosis of gut microbiota has been reported to be involved in the development of hypercholesterolemia in both humans and animal models. Probiotics have been reported to have ameliorative effects in murine models. However, whether probiotics could help alleviate dyslipidemia in adults remain obscure.

DETAILED DESCRIPTION:
Probiotics are live microorganisms that have been associated with multiple health benefits. However, its protective role in adults has long been controversial. This study aims to examine the effect of 12-week probiotics supplementation on lipid management in Chinese adults. By understanding the mechanism by which probiotics exert the beneficial effects, we can better control the rising prevalence of hypercholesterolemia, which is a major risk factor for cardiovascular diseases.

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects include men and women 18 to 75 years of age with primary hypercholesterolemia who has a total cholesterol level of 5.18 mmol/L or higher and/ or an LDL cholesterol level of 2.59 mmol/L or higher;
* Absence of any diet, dietary supplement and medication that might interfere with lipid homoeostasis and gut microbiota, especially antibiotics and probiotics.

Exclusion Criteria:

* Triglyceride levels higher than 3.95 mmol/L, or any other systemic, metabolic and cardiovascular or cerebrovascular diseases;
* Type 1 diabetes, type 2 diabetes treated with insulin or other medications;
* Acute illness or current evidence of acute or chronic inflammatory or infective diseases;
* Participation in any diet or lifestyle program more than 2 times per week in the latest 3 months prior to recruitment;
* Mental illness rendering them unable to understand the nature, scope, and possible consequences of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-05-12 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Total cholesterol | baseline, 4 weeks, 8 weeks and 12 weeks
  changes of total cholesterol levels in plasma by automatic biochemical analyzer
LDL-cholesterol | baseline, 4 weeks, 8 weeks and 12 weeks
  changes of LDL-cholesterol levels in plasma by automatic biochemical analyzer
Triglyceride | baseline, 4 weeks, 8 weeks and 12 weeks
  changes of triglyceride levels in plasma by automatic biochemical analyzer
non HDL-cholesterol | baseline, 4 weeks, 8 weeks and 12 weeks
  changes of non HDL-cholesterol levels in plasma
gut microbiota | baseline, 4 week, 8 weeks and 12 weeks
  changes of gut microbiota by metagenomics

SECONDARY OUTCOMES:
blood pressure | baseline, 4 week, 8 week and 12 weeks
  changes of blood pressure
pulse wave velocity | baseline and after 12-week intervention
  changes of pulse wave velocity by VP-1000plus from Omron
ankle Brachial Index | baseline and after 12-week intervention
  changes of ankle Brachial Index by VP-1000plus from Omron
microbial metabolite | baseline and after 12-week intervention
  changes of microbial metabolite by untargeted metabolomics

CONTACTS AND LOCATIONS:
Overall Officials: Min Xia, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Department of Nutrition and Food Hygiene, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No